CLINICAL TRIAL: NCT01016288
Title: Multicenter Randomized Controlled Trial Comparing the Performance of 22 Gauge Versus 25 Gauge EUS-FNA Needles
Brief Title: Controlled Trial Comparing the Performance of 22 Gauge Versus 25 Gauge EUS-FNA Needles (FNA-22G-25G)
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Medicine and Pharmacy Craiova (Other); Allgemeines Krankenhaus Celle, Celle, Germany (Unknown); Pathologic Institute, Wittinger Strasse, Celle, Germany (Unknown); Sana Hospital Lübeck GmbH, Lübeck, Germany (Unknown); LungenClinic Grosshansdorf (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Peter Vilmann, Professor, University Hospital, Gentofte, Copenhagen
Other Study IDs: EUS-FNA-DK-PV-2009
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Mediastinal Tumours and Lymph Nodes; Celiac, Perigastric and Peri-pancreatic Lymph Nodes; Pancreatic Masses; Liver Masses; Adrenal Masses
Keywords: EUS-FNA; 22 Gauge Needle; 25 Gauge Needle
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pathology samples obtained through EUS-FNA biopsy processed by paraffin embedding.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 22 G Needle EUS-FNA: Patients referred for an EUS examination and EUS-FNA of a solid mass lesion adjacent to the upper GI tract using a 22 G needle
- 25 G Needle EUS-FNA: Patients referred for an EUS examination and EUS-FNA of a solid mass lesion adjacent to the upper GI tract using a 25 G needle

SUMMARY:
The aim of the study is to compare the performance characteristics of EUS-FNA 22 Gauge needle and EUS FNA 25 Gauge needle in terms of cellularity and diagnostic yield for diagnosis of various pathologies, including lymph nodes, pancreatic, luminal and other lesions outlined by EUS.

DETAILED DESCRIPTION:
Tissue acquisition by Endoscopic ultrasound plays a central role in diagnosis of several pathologies; this is achieved by obtaining cytological material with fine needle aspiration (FNA) needles that are able to provide smears of malignant cells. Several needles are at present available including 19 Gauge, 22 Gauge and 25 Gauge needles. A 22 Gauge needle is at present the standard needle and most of the EUS-FNA results are based on FNA with this needle.

Twenty five Gauge needles presently available on the market are distinctly small, highly flexible and may be easier to penetrate hard pancreatic tumors. There even is anecdotal messages that this size of needle may be able to traverse relatively large vascular structures without major risk. However, there is very scant data on whether a 25 G needle is comparable to a standard 22 G needle in terms of specimen cellularity and quality. There is only one small randomized trial published as an abstract by Lee et al reporting no statistical significant difference in cellularity between the two groups of needle size as judged by 2 different cytologists. However, the conclusion is dubious because considerable bias may be present since both needles were used in the same lesion. There is therefore a need for a properly designed randomized study comparing different needle sizes.

This study is a prospective randomized multicenter study. Patients referred to one of the participating departments for an EUS examination will be included prospectively. Linear EUS examination will be done with a linear echoendoscope for lymph nodes, mediastinal, pancreatic and other intra-abdominal masses.

Tumor and lymph node characteristics will be carefully described: size (long axis), echogeneity (hypoechoic, hyperechoic, mixed), and echostructure (homogenous, in-homogenous, calcifications), shape (round, oval, triangular), border (regular, irregular).

EUS-guided cell sampling will be performed with a 22 G (Medi-Globe, Sonotip II) and 25 G (Medi-Globe, Sonotip II) needles under EUS and Colour-Doppler guidance.

Needle order will be selected randomly, one single needle pr. Lesion. Three passes will be performed with either of the needles after randomization, using 6 uniform to and fro movements on every pass with continuous 10cc suction for the reason of standardization. The material will be expelled on separate numbered glass slides. The cytopathologist will review the material after staining blinded to the needle size and will be using standardized criteria for evaluation of cellularity.

Doubtless, this multicenter randomized controlled trial comparison, as any other experimental method, needs with necessity a serious statistical evaluation, bringing the benefits of improving the reliability and credibility of the findings thus obtained. Accordingly, both exploratory data analysis and statistical inference will be performed. Technically, the expected number of lesions to be included in the study will be 220, 110 in each group. Block randomization (block size = 4) will be used to ensure exactly equal treatment numbers at certain equally spaced points in the sequence of patients assignments (Knuth shuffle algorithm for random permutations).

For diagnostic tests the sensitivity, specificity positive and negative predictive value and diagnostic accuracy will be calculated and calculated separately for EUS-FNA during 1st pass, 2nd pass and 3rd pass by comparing the results with the final diagnosis. All results will be expressed as mean, standard deviation (SD) and confidence interval. Testing hypotheses will be used afterwards. An a priori power analysis will be performed to determine the appropriate sample size in order to achieve adequate power for the statistical tests subsequently used. The data from both groups will be compared by standard comparison tests chi-square test or Fishers exact test where appropriate. The level of statistical significance is stated as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for an EUS examination and EUS-FNA of a solid mass lesion adjacent to the upper GI tract
* Well informed signed consent for EUS-guided FNA

Exclusion Criteria:

* Severe coagulopathy
* Uncorrectable severe platelet dysfunction
* Presence of large intervening vessels on color or power Doppler
* Failure to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to one of the participating departments for an EUS examination with EUS-FNA (mediastinal tumours and lymph nodes, celiac, perigastric and peri-pancreatic lymph nodes, pancreatic masses, liver masses, adrenal masses, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Value of EUS-FNA 22 Gauge needle comparing with EUS-FNA 25 Gauge needle in terms of cellularity and diagnostic yield for diagnosis of various pathologies. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vilmann, Professor, Study Director — Gentofte Hospital, Copenhagen University, Denmark
Locations (9):
- Denmark (2):
  - Department of Pathology, Herlev University Hospital, Hellerup, Copenhagen
  - Endoscopy Z-806, Gentofte, Department of Surgical Gastroenterology, Gentofte and Herlev Hospitals, Copenhagen
- Germany (6):
  - Department of Medicine, GI Division, Allgemeines Krankenhaus MD, Celle
  - Klinik für Gastroenterologie/GI-Onkologie, Allgemeines Krankenhaus Celle, Celle
  - Pathologic Institute, Wittinger Strasse, Celle
  - Cytological Laboratory, Hospital Grosshansdorf - Center for Pneumology and Thoracic Surgery, Großhansdorf
  - Department of Internal Medicine, Sana Hospital Lübeck GmbHg, MD, Lübeck
  - Department of Pathology, Medical University Schleswig-Holstein, Lübeck
- Research Center of Gastroenterology and Hepatology, University of Medicine and Pharmacy, Craiova, Romania

REFERENCES:
- [Background] Vilmann P, Puri R. The complete ''medical'' mediastinoscopy (EUS-FNA + EBUS-TBNA). Minerva Med. 2007 Aug;98(4):331-8. PMID 17921946
- [Background] Saftoiu A, Vilmann P, Guldhammer Skov B, Georgescu CV. Endoscopic ultrasound (EUS)-guided Trucut biopsy adds significant information to EUS-guided fine-needle aspiration in selected patients: a prospective study. Scand J Gastroenterol. 2007 Jan;42(1):117-25. doi: 10.1080/00365520600789800. PMID 17190771
- [Derived] Vilmann P, Saftoiu A, Hollerbach S, Skov BG, Linnemann D, Popescu CF, Wellmann A, Gorunescu F, Clementsen P, Freund U, Flemming P, Hassan H, Gheonea DI, Streba L, Ioncica AM, Streba CT. Multicenter randomized controlled trial comparing the performance of 22 gauge versus 25 gauge EUS-FNA needles in solid masses. Scand J Gastroenterol. 2013 Jul;48(7):877-83. doi: 10.3109/00365521.2013.799222. PMID 23795663